CLINICAL TRIAL: NCT05464147
Title: DYNAMX Bioadaptor ImplanTation for the trEatment of Complex Coronary Lesions (DYNAMITE Study)
Brief Title: DYNAMX Bioadaptor ImplanTation for the trEatment of Complex Coronary Lesions
Acronym: DYNAMITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Elixir Medical Corporation (Industry)
Collaborators: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Dr. Antonio Colombo, Dr. Antionio Colombo, Senior Consultant - Cardio Center, Clinical and Interventional Cardiology Unit, IRCCS Humanitas Research Hospital, Rozzano, Italy, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 250521
Record Dates: First submitted 2022-07-13; First posted 2022-07-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease; Chronic Total Occlusion of Coronary Artery; Bifurcation of Coronary Artery; Multi Vessel Coronary Artery Disease; Long Lesions Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Masking Description: All imaging analyses will be performed at an independent core laboratory (Cardiovascular Department, San Giovanni Addolorata Hospital, Rome, Italy) by experienced operators blinded to procedural data and clinical outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- DynamX Drug-Eluting Coronary Bioadaptor System (Experimental)
  Interventions: Device: DynamX Drug-Eluting Coronary Bioadaptor System

INTERVENTIONS:
Device: DynamX Drug-Eluting Coronary Bioadaptor System — DynamX Drug-Eluting Coronary Bioadaptor System Implantation in Coronary Artery Lesion

SUMMARY:
The aim of the DYNAMITE study is to investigate the (a) acute procedural and (b) 9-month follow-up performance of DynamX Drug-Eluting Coronary Bioadaptor System implantation in complex coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

Presence of complex coronary lesions defined as follows:

* long lesions (>28 mm);
* CTO, a total occlusion of duration more than 3-months;
* Lesions involving a bifurcation, defined as a division with a side branch large enough to be stented (i.e. >2.25 mm);
* Patients requiring 4 or more stents
* Reference vessel diameter: >2.25 mm to <4.0 mm

Exclusion Criteria:

* Age under 18 years old;
* Significant co-morbidity precluding clinical follow-up;
* A positive pregnancy test in women with child-bearing potential;
* Contra-indication to dual anti-platelet therapy;
* Thrombocytopenia <100,000/uL;
* Major surgery planned which will lead to discontinuation of antiplatelet therapy;
* In-stent restenosis;
* Treatment of saphenous vein graft;
* CTO with long sub-intimal tracking (> 20 mm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in mean in-device lumen area and mean device area | Through 9 months
  Change in mean in-device lumen area and mean device area, as measured by Optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Major Adverse Cardiac Event (MACE) | 9 months, 12 months and 24 months
  Major adverse cardiac event (MACE) (composite of cardiac death, myocardial infarction [MI], and target lesion revascularization [TLR])
Cardiac Death (CD) | 9 months, 12 months and 24 months
  Cardiac Death (CD)
Myocardial Infarction (MI) | 9 months, 12 months and 24 months
  Myocardial Infarction (MI)
Target Lesion Revascularization (TLR) | 9 months, 12 months and 24 months
  Target Lesion Revascularization (TLR)
Stent Thrombosis (ST) | 9 months, 12 months and 24 months
  Stent Thrombosis (ST)
Stent Cross-Sectional Area | 9 months
  Stent Cross-Sectional Area by OCT
Minimum stent diameter | 9 months
  Minimum stent diameter by OCT
Maximum stent diameter | 9 months
  Maximum stent diameter by OCT
Intimal hyperplasia (IH) area | 9 months
  Intimal hyperplasia (IH) area (calculated as stent area minus luminal area) by OCT
Percentage of intimal hyperplasia | 9 months
  Percentage of intimal hyperplasia (IH area divided by stent area) by OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Italy